CLINICAL TRIAL: NCT02995278
Title: Clinical Researcher Experience Assessment Documenting Usage and Plan of Care Changes Due to Drug Screenings ©
Brief Title: Usage and Plan of Care Changes Due to Drug Screenings
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Data Collection Analysis Business Management (Other)
Collaborators: PAS Research Services (Other)
Responsible Party: Sponsor
Other Study IDs: PAS1459
Record Dates: First submitted 2016-12-06; First posted 2016-12-16 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Does not include a drug needing FDA approval and therefore it is not by definition, a Clinical Drug Trial as defined by FDA.

SUMMARY:
The purpose of this minimal risk, observational survey is to document the accuracy, benefits, and how qualitative and quantitative results affect patients' plan of care.

DETAILED DESCRIPTION:
Pain is the most common reason patients consult primary care providers. According to recent surveys, One in six Americans live with chronic or recurrent pain and pay an estimated $120 billion a year in medical costs in the United States. Oral opioids are the common treatment options for various chronic pains including joint pain, musculoskeletal pain, neuropathic pain and migraines. This narcotic-based management of pain is often associated with undesirable side effects with addictive and potential abuse.

To ensure proper usage of prescribed medications, physicians use drug screens to monitor therapeutic levels and test for presence of illegal drugs or medications that may cause a drug-drug interaction. Upon receiving quantitative or qualitative results from these drug screens, the physician may change the treatment plan for patients to improve efficacy of prescribed medications.

ELIGIBILITY:
Inclusion Criteria:

* Must be a Medical Practioner

  * Medical Doctor (MD)
  * Doctor of Osteopathic (DO)
  * Physician Assistant (PA)
  * Advanced Practice Registered Nurse (APRN)
  * Nurse Practioner (NP)
* Must have a current standard operating procedure that includes obtaining/reviewing medical history.

Exclusion Criteria:

* Government-funded insurance data cannot be included in the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Providers who already drug screen for their current patient population.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Plan of Care Changes due to Drug Screenings | 3 years
  Provider based observational survey

IPD SHARING:
Plan to Share IPD: Undecided
Plan of care changes by providers after toxicology testing